CLINICAL TRIAL: NCT05025800
Title: A Phase I/II Open Label, Single Center, Study of the Combination of ALX148, Rituximab and Lenalidomide in Patients With Indolent and Aggressive B-Cell Non-Hodgkin Lymphoma
Brief Title: ALX148, Rituximab and Lenalidomide for the Treatment of Indolent and Aggressive B-cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0226; NCI-2021-08492 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0226 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-05; First posted 2021-08-27 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Aggressive B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage III Grade 3 Follicular Lymphoma; Ann Arbor Stage III Marginal Zone Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Grade 3 Follicular Lymphoma; Ann Arbor Stage IV Marginal Zone Lymphoma; Composite Lymphoma; Indolent B-Cell Non-Hodgkin Lymphoma; Refractory Aggressive B-Cell Non-Hodgkin Lymphoma; Refractory Follicular Lymphoma; Refractory Grade 3b Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Transformed Marginal Zone Lymphoma to Diffuse Large B-Cell Lymphoma; Richter Syndrome
MeSH Terms: conditions — Composite Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — ALX148; Lenalidomide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ALX148, rituximab, lenalidomide) (Experimental): Patients receive ALX148 IV over 1 hour once on days 1, 8, 15 and 22, or days 1 and 15, or day 1 depending on dose level. Patients also receive rituximab IV over 4-6 hours on days 1, 8, 15 and 22 of cycle 1, then on day 1 of cycles 2-6, and lenalidomide PO QD on days 1-21 of cycles 1-6. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: CD47 Antagonist ALX148; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: CD47 Antagonist ALX148 — Given IV
  Other Names: ALX 148; ALX-148; ALX148; CD47/SIRPa-blocking Agent ALX148; SIRPa Variant ALX148
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase I/II trial finds out the best dose, possible benefits and/or side effects of ALX148 in combination with rituximab and lenalidomide in treating patients with indolent and aggressive B-cell non-Hodgkin lymphoma. Immunotherapy with ALX148, may induce changes in body's immune system and may interfere with the ability of cancer cells to grow and spread. Chemotherapy drugs, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Rituximab is a monoclonal antibody that binds to a protein called CD20 found on B-cells, and may kill cancer cells. Giving ALX148 in combination with rituximab and lenalidomide may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate safety and tolerability, and to determine the recommended phase II dose (RP2D) and schedule of CD47 antagonist ALX148 (ALX148) in combination with rituximab and lenalidomide in patients with relapsed or refractory B-non-Hodgkin lymphomas (NHLs) (both indolent and aggressive histology) in phase I.

II. To evaluate the efficacy of the combination of ALX148, rituximab and lenalidomide at the RP2D (determined in phase I) in patients with previously untreated and high tumor burden indolent B-NHL in phase II.

SECONDARY OBJECTIVE:

I. To evaluate other toxicity and efficacy measures of the combination of ALX148, rituximab and lenalidomide.

EXPLORATORY OBJECTIVE:

I. To determine the pharmacodynamic effects and investigate biomarkers of response and resistance.

OUTLINE: This is a phase I, dose-escalation study of ALX148 followed by a phase II study.

Patients receive ALX148 intravenously (IV) over 1 hour once on days 1, 8, 15 and 22, or days 1 and 15, or day 1 depending on dose level. Patients also receive rituximab IV over 4-6 hours on days 1, 8, 15 and 22 of cycle 1, then on day 1 of cycles 2-6, and lenalidomide orally (PO) daily once (QD) on days 1-21 of cycles 1-6. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 7 and 30 days, then up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: histologically confirmed B-cell NHL, including marginal zone lymphoma, follicular lymphoma, mantle cell lymphoma, large B-cell lymphoma (including transformed MZL, transformed FL, Richter Syndrome with ALC < 5,000 109/L, FL grade 3B, high grade B-cell lymphoma and primary mediastinal B-cell lymphoma), and composite lymphoma (concomitant indolent and aggressive B-NHL)
* Phase I: have failed at least one line of systemic therapy and not be eligible for known standard of care curative treatment option; patients with mantle cell lymphoma and aggressive B-cell lymphoma will need to have received 2 prior lines of systemic therapy.
* Phase II: histologically confirmed follicular lymphoma, grade 1, 2, or 3a or marginal zone lymphoma
* Phase II: have had no prior systemic treatment for lymphoma
* Phase II: high tumor burden disease, defined by meeting 1 or more of the following GELF criteria

  * Bulky disease defined as: a nodal or extranodal (except spleen) mass >7cm in its greater diameter or, involvement of at least 3 nodal or extranodal sites (each with a diameter greater than >3 cm)
  * Presence of at least one of the following B symptoms: fever (>38C) of unclear etiology, night sweats, weight loss greater than 10% within the prior 6 months
  * Symptomatic splenomegaly
  * Impending organ compression or involvement
  * Any one of the following cytopenias due to lymphoma: hemoglobin < 10 g/dL (6.25 mmol/L), platelets < 100 x 10^9/L , or absolute neutrophil count (ANC) < 1.5 x 10^9 /L
  * Pleural or peritoneal serous effusion (irrespective of cell content)
  * Lactate dehydrogenase [LDH] > upper limit of normal (ULN) or beta 2 microglobulin > ULN
* Phase II: stage III or IV disease
* Bi-dimensionally measurable disease, with at least one nodal lesion >= 1.5 cm or one extra-nodal lesion >= 1 cm in longest diameter by computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI)
* Must be >= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) >= 1,000/mm^3, independent of growth factor support (within 28 days prior to signing informed consent)
* Platelet counts >= 75,000/mm^3 or >= 50,000/mm^3 if bone marrow involvement with lymphoma, independent of transfusion support for >= 14 days in either situation (within 28 days prior to signing informed consent)
* Hemoglobin > 8 g/dL, independent of transfusion support for >= 14 days (within 28 days prior to signing informed consent)
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) < 2 x upper limit of normal (ULN)
* Creatinine clearance > 30 ml/min calculated by modified Cockcroft-Gault formula
* Total bilirubin < 1.5 x ULN unless bilirubin is due to Gilbert's syndrome, documented liver involvement with lymphoma, or of non-hepatic origin, in which case bilirubin should not exceed 3 g/dL
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) < 1.5 x ULN
* Must be able to adhere to the study visit schedule and other protocol requirements
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study (females of childbearing potential: must either completely abstain from heterosexual sexual conduct or must use 2 methods of reliable contraception, 1 highly effective [intrauterine device, birth control pills, hormonal patches, injections, vaginal rings, or implants] and at least 1 additional method [condom, diaphragm, cervical cap] of birth control). Reliable contraceptive methods must be started at least 4 weeks before lenalidomide, and continued for at least 4 weeks after last dose of lenalidomide. Males who are sexually active must be practicing complete abstinence or agree to a condom during sexual contact with a pregnant female or female of child bearing potential. Men must agree to not donate sperm during the study and 28 days after the last dose of lenalidomide. For females, these restrictions apply at least 4 weeks before study treatment, during the period of therapy and for 120 days after the last dose of study drug. For males, these restrictions apply during the period of therapy and for 28 days after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study.

  * Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program

Exclusion Criteria:

* Known active central nervous system lymphoma or leptomeningeal disease, except subjects with a history of central nervous system lymphoma treated and in remission > 6 months
* Burkitt lymphoma
* Chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) or lymphoplasmacytic lymphoma (LPL)/Waldenstrom macroglobulinemia
* Any prior history of other malignancy besides B-NHL, unless the patient has been free of disease for >= 3 years and felt to be at low risk for recurrence by the treating physician, except:

  * Adequately treated localized skin cancer without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of lenalidomide capsules, or put the study outcomes at undue risk
* Known history of human immunodeficiency virus (HIV), or active hepatitis C virus, or active hepatitis B virus infection, or any uncontrolled active significant infection, including suspected or confirmed JC virus infection and severe acute respiratory syndrome coronavirus 2 (SARS-CoV2)

  * Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of hepatitis C who received antiviral treatment are eligible as long as PCR is negative
* History of immunodeficiency (with the exception of hypogammaglobulinemia) or concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of > 10 mg/day of prednisone) within 28 days of the first dose of study drug
* Known anaphylaxis or immunoglobulin (Ig)E-mediated hypersensitivity to murine proteins or to any component of ALX148, lenalidomide and/or rituximab.

  * In regards to rituximab, exclusion is for known severe anaphylaxis to rituximab or any allergic reaction to rituximab that in the opinion of the PI and treating physician contraindicate re-challenge with rituximab
* Requires chronic treatment with strong CYP3A inhibitors, for a list of strong CYP3A inhibitors. If patients have been on a strong CYP3A inhibitor in the past, they will not be eligible if the CYP3A inhibitor was administered within 7 days of the first dose of study drug
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block
* Active bleeding or known bleeding diathesis (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to study entry
* Vaccinated with live, attenuated vaccines within 4 weeks of study entry
* Lactating or pregnant subjects
* Administration of any investigational agent within 28 days of first dose of study drug
* Patients who have undergone major surgery within 28 days or minor surgery within 3 days of first dose of study drug
* Patients taking corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 10 mg/day prednisone (over these 4 weeks)
* Life expectancy < 6 months
* Neuropathy > grade 1
* Prior exposure to lenalidomide or to a CD47/SIRP alpha antagonist/inhibitor, independently from indication
* Patient who received chimeric antigen receptor (CAR) T-cell therapy within 1 month, autologous stem cell transplant within 3 months, allogeneic stem cell transplant within 6 months
* Patients who have difficulty with or are unable to swallow oral medication, or have disease significantly affecting gastrointestinal function that would limit absorption of oral medication
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
* History of hemolytic transfusion reaction secondary to allo-antibodies
* Patients who have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed. Agents with limited immunosuppressive activity (ex. Hydroxychloroquine) are allowed after discussion with the study PI ).
* Patients who have a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Known history of symptomatic deep vein thrombosis or pulmonary embolism
* Known history of Stevens-Johnson syndrome (SJS) or toxic epidermal necrolysis (TEN) or drug rash with eosinophilia and systemic symptoms (DRESS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) and schedule of ALX148 (Phase I) | Up to 28 days
Complete remission (CR) rate (Phase II) | At 6 months
  Response will be assessed by the investigator based on the 2014 Cheson Lugano criteria. The number and percentage of subjects with a CR at the end of treatment will be tabulated. The CR rate will be estimated with its exact 95% confidence interval (CI).

SECONDARY OUTCOMES:
Overall response rate (ORR) (CR + partial response [PR]) | After 6 cycles of treatment (At the end of Cycle 1 (each cycle is 28 days)
  Will be assessed by the investigator based on Cheson, Lugano 2014. The number and percentage of subjects with an ORR will be tabulated. The best ORR will be recorded and summarized using exact method for 95% CI.
Duration of response | From the time by which measurement criteria for CR or PR, whichever is recorded first, is met until death or the first date by which progressive disease is documented, assessed up to 3 years
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Progression-free survival (PFS) | From the date of cycle 1, day 1 (At the end of Cycle 1 (each cycle is 28 days)
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Overall survival (OS) | From the date of cycle 1, day 1 (At the end of Cycle 1 (each cycle is 28 days)
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Incidence of treatment-emergent adverse events (AEs) | Up to 30 days
  Safety summaries will include tabulations in the form of tables and listings. The frequency (number and percentage) of treatment-emergent AEs will be reported. Additional AE summaries will include AE frequency by AE severity and by relationship to study drug. Clinically significant abnormal laboratory values will be summarized.
Incidence of treatment-emergent AEs requiring temporary or permanent discontinuation of study drug or dose reductions | Up to 30 days
  Safety summaries will include tabulations in the form of tables and listings. The frequency (number and percentage) of treatment-emergent AEs will be reported. Additional AE summaries will include AE frequency by AE severity and by relationship to study drug. Clinically significant abnormal laboratory values will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Strati, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org